CLINICAL TRIAL: NCT00006454
Title: Phase III Multicenter Study in Epithelial Ovarian Carcinoma FIGO Stage IIB-IV Comparing Treatment With Paclitaxel and Carboplatin to Paclitaxel and Carboplatin Sequentially Followed by Topotecan
Brief Title: Paclitaxel Plus Carboplatin With or Without Topotecan in Treating Patients With Stage IIB, Stage III, or Stage IV Ovarian Epithelial Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AGO Study Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000067994; AGOSG-OVAR-7; NCI-V00-1602
Record Dates: First submitted 2000-11-06; First posted 2004-02-03 (Estimated); Last update posted 2015-12-23 (Estimated); Status verified 2015-12

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer
Keywords: stage II ovarian epithelial cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; fallopian tube cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Carboplatin; Paclitaxel; Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: carboplatin
Drug: paclitaxel
Drug: topotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. It is not yet known if paclitaxel plus carboplatin is more effective with or without topotecan for ovarian epithelial cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of paclitaxel plus carboplatin with or without topotecan in treating patients who have stage IIB, stage III, or stage IV ovarian epithelial cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare survival of patients with stage IIB, III, or IV ovarian epithelial carcinoma after receiving treatment with paclitaxel and carboplatin with or without topotecan. II. Compare progression-free survival of these patients after receiving these treatment regimens. III. Compare the response rate and response duration in these patients treated with these regimens. IV. Determine the toxic effects of the combination of paclitaxel, carboplatin, and topotecan in these patients. V. Compare the toxic effects of these treatment regimens in these patients. VI. Compare quality of life of these patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to participating center and stage (stage IIB and stage III optimally debulked to no greater than 1 cm residual tumor vs stage IV regardless of residual tumor or residual tumor greater than 1 cm). Patients are randomized to one of two treatment arms. Arm I: Patients receive paclitaxel IV over 3 hours and carboplatin IV over 0.5-1 hour on day 1 and topotecan IV over 0.5 hour on days 1-5. Treatment repeats every 21 days for 6 courses (topotecan is administered for 4 courses only). Arm II: Patients receive paclitaxel and carboplatin as in arm I. Treatment repeats every 21 days for 6 courses. Quality of life is assessed before courses 1, 3, and 5 and at 3 weeks and 3 months after completion of treatment in both treatment arms; before courses 1 and 3 of topotecan in arm I; and at 6 months after completion of treatment in arm II. Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 914 patients (457 per treatment arm) will be accrued for this study over 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed stage IIB, III, or IV ovarian epithelial carcinoma, fallopian tube, or extraovarian papillary serous carcinoma extending to the ovary No mixed epithelial/non-epithelial tumors (e.g., mixed Mullerian tumors) No tumors of low malignant potential (e.g., borderline tumors) No symptomatic brain metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 OR Karnofsky 70-100% Life expectancy: More than 12 weeks Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 times the upper limit of normal (ULN) Alkaline phosphatase no greater than 3 times ULN Renal: Creatinine no greater than 1.25 times ULN Estimated glomerular filtration rate at least 60 mL/min Cardiovascular: No history of congestive heart failure (even if medically controlled) No New York Heart Association class III or IV heart disease No myocardial infarction within the past 6 months No history of atrial or ventricular arrhythmias Other: No motor or sensory neurologic pathology or symptoms greater than grade 1 No active infection or other serious medical condition that would preclude study No prior allergy to drug containing Cremophor EL No dementia or significantly altered mental state that would preclude informed consent No complete bowel obstruction No other prior malignancy except curatively treated nonmelanomatous skin cancer or carcinoma in situ of the cervix Not pregnant or nursing Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent immunotherapy No concurrent WBC transfusions Chemotherapy: No prior chemotherapy No other concurrent chemotherapy Endocrine therapy: No concurrent hormonal therapy Radiotherapy: No prior radiotherapy No concurrent radiotherapy Surgery: No more than 6 weeks since prior definitive laparotomy and recovered Other: No other concurrent antineoplastic agents No other concurrent investigational drugs

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-12; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacobus Pfisterer, MD, Study Chair — University Hospital Schleswig-Holstein
Locations (19):
- Germany (19):
  - Universitaetsklinikum Charite, Berlin
  - Universitaetskliniken Bonn, Bonn
  - Zentralkrankenhaus, Bremen
  - Medizinische Klinik I, Dresden
  - Universitaetsklinik Duesseldorf, Düsseldorf
  - Evangelisches Krankenhaus, Düsseldorf
  - Klinikum der J.W. Goethe Universitaet, Frankfurt
  - Stadtische Kliniken Frankfurt-Hochst, Frankfurt
  - Universitaetsklinik Goettingen, Göttingen
  - Klinik Fuer Innere Medizin Hematology/Oncology, Ernst Moritz Armdt Universitaet, Greifswald
  - Frauenklinik der MHH, Hanover
  - Vincentius Krankenhaus, Karlsruhe
  - Christian-Albrechts University of Kiel, Kiel
  - Klinik der Otto-v.-Guericke-Universitat, Magdeburg
  - Klinikum Grosshadern, Munich
  - Klinikum Rechts Der Isar/Technische Universitaet Muenchen, Munich
  - Klinik und Poliklinik fuer Kinderheilkunde, Münster
  - Universitaetsklinikum Tuebingen, Tübingen
  - Dr. Horst-Schmidt-Kliniken, Wiesbaden

REFERENCES:
- [Background] Greimel ER, Bjelic-Radisic V, Pfisterer J, Hilpert F, Daghofer F, Pujade-Lauraine E, du Bois A; Arbeitsgemeinschaft Gynaekologische Onkologie Ovarian Cancer Study Group (AGO-OVAR); Groupe d'Investigateurs Nationaux pour les Etudes des Cancers de l'Ovaire (GINECO). Toxicity and quality of life outcomes in ovarian cancer patients participating in randomized controlled trials. Support Care Cancer. 2011 Sep;19(9):1421-7. doi: 10.1007/s00520-010-0969-8. Epub 2010 Aug 6. PMID 20694564
- [Result] Pfisterer J, Weber B, Reuss A, Kimmig R, du Bois A, Wagner U, Bourgeois H, Meier W, Costa S, Blohmer JU, Lortholary A, Olbricht S, Stahle A, Jackisch C, Hardy-Bessard AC, Mobus V, Quaas J, Richter B, Schroder W, Geay JF, Luck HJ, Kuhn W, Meden H, Nitz U, Pujade-Lauraine E; AGO-OVAR; GINECO. Randomized phase III trial of topotecan following carboplatin and paclitaxel in first-line treatment of advanced ovarian cancer: a gynecologic cancer intergroup trial of the AGO-OVAR and GINECO. J Natl Cancer Inst. 2006 Aug 2;98(15):1036-45. doi: 10.1093/jnci/djj296. PMID 16882940
- [Result] Pfisterer J, Lortholary A, Kimmig R, et al.: Paclitaxel/carboplatin (TC) vs. paclitaxel/carboplatin followed by topotecan (TC-Top) in first-line treatment of ovarian cancer FIGO stages IIb - IV. Interim results of a gynecologic cancer intergroup phase III trial of the AGO Ovarian Cancer Study Group and GINECO. [Abstract] Proceedings of the American Society of Clinical Oncology 22: A-1793, 446, 2003.